CLINICAL TRIAL: NCT06157879
Title: Measuring Electrical Properties of Breast Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Wave View Imaging (Unknown); Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HREBA.CC-22-0112
Record Dates: First submitted 2023-11-06; First posted 2023-12-06 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Breast
Keywords: women

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- WVI-MIS-01-2022 (Experimental): Healthy volunteers
  Interventions: Device: WVI-MIS-01-2022

INTERVENTIONS:
Device: WVI-MIS-01-2022 — Microwave scans

SUMMARY:
The goal of this observational study is to use a low-powered microwave imaging system to provide insight into the correlation of electrical properties of breast tissue at microwave frequencies and breast density obtained from mammograms in healthy women between the ages of 18 and 74. The main questions it aims to answer : • Is there a correlation between the electrical properties of breast tissue and breast density obtained from mammograms? Both breasts of each participant will be scanned by the microwave imaging system six times in total.

DETAILED DESCRIPTION:
A new approach to imaging that uses low-power microwaves to scan the breast has been developed. Since the imaging system uses low power, there is no risk of tissue heating. The imaging system places the sensors in contact with the breast and does not require compression. The research team at the University of Calgary has previously developed microwave imaging systems that have been tested on volunteers and patients. This included repeated scanning of a group of volunteers to evaluate the consistency of the approach. The information collected from experiences scanning volunteers and patients have been reviewed and translated into a next-generation imaging system design. Aspects of this system have been further improved by Wave View Imaging, which is a company formed by members of the University's research team.

The proposed study involves collecting electrical property measurements of breast tissues and comparing these measurements to clinical information. The investigators also aim to compare regions of interest in the microwave scans with regions of interest in the mammograms. This includes regions dominated by fibroglandular tissues, as well as regions of interest that correspond to anomalies identified in the mammograms

The plan is to scan both breasts of up to 200 volunteers. Each volunteer will participate in a single scanning session. Breast tissue composition (VOLPARA score) will be compared with the microwave properties and registration of mammograms with microwave images will be performed for a more detailed comparison.

ELIGIBILITY:
Inclusion Criteria:

* Must have had a previous mammogram in the last 2 years

Exclusion Criteria:

* Participants currently undergoing chemotherapy and/or radiation treatment.
* Participants with breast implants.
* Participants who are breast or breastfeeding.
* Participants with active breast infections.
* Participants with nipple piercings (unless they can be removed prior to scanning).
* Participants with an implanted electronic device.
* Participants with physical limitations that prevent them from placing their breasts in the scanner.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Measurement of electrical properties of breast tissue | 18 months
  The electrical properties will be estimated for each volunteer and an image that maps these properties will be created.

SECONDARY OUTCOMES:
Correlation between the electrical properties of breast tissue and breast density | 18 months
  Comparison of the microwave images and mammograms in 2 ways: VOLPARA scores versus average electrical properties and comparison of regions of interest in both images

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith, K., et al. "Microwave Imaging of the Breast: Consistency of Measurements Over Time." IEEE Journal of Electromagnetics, RF and Microwaves in Medicine and Biology, vol. 6, no. 1, 2022, pp. 61-67, https://doi.org/10.1109/JERM.2021.3099014.
- [Background] Smith K, Bourqui J, Wang Z, Besler B, Lesiuk M, Roumeliotis M, Quirk S, Grendarova P, Pinilla J, Price S, Docktor B, Fear E. Microwave imaging for monitoring breast cancer treatment: A pilot study. Med Phys. 2023 Nov;50(11):7118-7129. doi: 10.1002/mp.16756. Epub 2023 Oct 6. PMID 37800880